CLINICAL TRIAL: NCT04791761
Title: Use of a Non-Opioid Pain Regimen for Post-Operative Analgesia Following Intracapsular Adenotonsillectomy
Brief Title: Non-Opioid Pain Medications After Intracapsular Adenotonsillectomy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: David Chi, MD (Other)
Responsible Party: Sponsor-Investigator, David Chi, MD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19040036 (Part 2)
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Results first posted 2024-08-16 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Adenotonsillectomy; Post-operative Analgesia; Opioid Use
Keywords: analgesia; pain control; adenotonsillectomy; tonsillectomy; opioids; post-operative pain; intracapsular
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Oxycodone; Ibuprofen; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Experimental, open-label randomized control trial.
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Opioid pain control (Experimental): Patients in this group will be receiving triple therapy for pain control with oxycodone, acetaminophen, and ibuprofen. They will be asked to complete a pain diary which will be used to determine the level of pain control achieved with this regimen. The diary will be completed by post-operative day 14. A post-operative appointment between 4-8 weeks will be scheduled and the patient and caregiver will return the pain diary or by email/mail if no appointment was scheduled. Families will receive an opioid disposal education document.
  Interventions: Drug: Oxycodone; Drug: Ibuprofen; Drug: Acetaminophen; Other: Opioid disposal education
- Opioid pain control + Disposal Pouch (Experimental): Patients in this group will be receiving triple therapy for pain control with oxycodone, acetaminophen, and ibuprofen. They will be asked to complete a pain diary which will be used to determine the level of pain control achieved with this regimen. The diary will be completed by post-operative day 14. A post-operative appointment between 4-8 weeks will be scheduled and the patient and caregiver will return the pain diary or by email/mail if no appointment was scheduled. Half of the families randomized to the opioid group will be further randomized to receive an opioid disposal bag + an opioid disposal education document. The pouch is a drug deactivation disposal pouch to dispose the opioid at home.
  Interventions: Drug: Oxycodone; Drug: Ibuprofen; Drug: Acetaminophen; Other: Opioid disposal pouch; Other: Opioid disposal education
- Non-opioid pain control (Active Comparator): Patients in this group will be receiving therapy for pain control with acetaminophen and ibuprofen only. They will be asked to complete a pain diary which will be used to determine the level of pain control achieved with this regimen. The diary will be completed by post-operative day 14. A post-operative appointment between 4-8 weeks will be scheduled and the patient and caregiver will return the diary or by email/mail if no appointment was scheduled.
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen

INTERVENTIONS:
Drug: Oxycodone — Oxycodone will be prescribed at a dose in the range of 0.025 mg/kg to 0.10 mg/kg every four hours or as needed for adequate pain management. The total supply will be limited to seven days. It will be prescribed in liquid suspension form for ease of use in pediatric populations. Subjects or parents will purchase this medication and dosage will be given to subjects in easy-to-understand language.
  Arms: Opioid pain control; Opioid pain control + Disposal Pouch
Drug: Ibuprofen — Ibuprofen will be prescribed at 10 mg/kg to be taken every 6 hours for the first three post-operative days. After the first three days, the subject should take the ibuprofen every 6 hours as needed for pain control. The daily dose of ibuprofen is not to exceed 1200mg or more than 4 individual doses. It will be prescribed in liquid suspension form for ease of use in pediatric populations. Subjects or parents will purchase this medication and dosage will be given to subjects in easy-to-understand language.
Drug: Acetaminophen — Acetaminophen will be prescribed at 15mg/kg to be taken every 4 hours for the first three days, except when sleeping. After the first three days, the subject should take the acetaminophen every 4 hours as needed for pain control. The daily dose of acetaminophen is not to exceed 5 doses in 24 hours. It will be prescribed in liquid suspension form for ease of use in pediatric populations. Subjects or parents will purchase this medication and dosage will be given to subjects in easy-to-understand language.
Other: Opioid disposal pouch — Half of the opioid group will be randomized assigned to an opioid disposal pouch arm. This pouch is a drug deactivation system that can be disposed in the trash in a household.
  Arms: Opioid pain control + Disposal Pouch
Other: Opioid disposal education — An opioid disposal education document will be provided to all families in the opioid group. This education document has information on unused or expired prescription medication disposal and specific information about permanent collection sites within our health system, drug take-back locations, drug take back day, and disposing at home.
  Arms: Opioid pain control; Opioid pain control + Disposal Pouch

SUMMARY:
The goal of this study is to determine if non-opioid pain control is a safe way to manage pain after intracapsular adenotonsillectomy surgery in children. This study is the second part of our randomized clinical trials of assessing pain after adenotonsillectomy (T&A), the first being total T&A. The investigators will repeat the methodology in the first clinical trial by randomly assigning children aged 3-17 to one of two groups: one group will receive non-opioid pain medication only, and the other group will receive opioid and non-opioid medications for pain control. The investigators will analyze the data and determine if there is a difference in pain control between the two drug regimens, and if there are any other associated complications between the two groups.

This study is important because if we can demonstrate that there is little difference in outcomes and pain control between the two groups, a strong argument can be made for reducing or eliminating opioid prescription after intracapsular adenotonsillectomy. This may protect future children from the risks of taking opioid medications and help to reduce the scope of the opioid epidemic.

DETAILED DESCRIPTION:
Purpose: To determine if non-opioid pain control is a safe and effective option in the treatment of post-operative pain following intracapsular adenotonsillectomy in various pediatric age groups.

Methods: The subject population will be patients between the ages of 3 and 17 who will undergo intracapsular adenotonsillectomy (T&A). Intracapsular versus total T&A technique will be predetermined by the child's physician and will not be a part of the study. The study will consist of two unblinded arms - patients receiving standard pain control regimen which include opioids and non-opioids, and patients receiving non-opioid pain medications only. In the diary they will receive, patients or caregivers will record frequency of pain medication taken each day with daily symptoms, a survey, and pain ratings measured by the Wong-Baker FACES Pain Rating Scale. Within 4-8 weeks post-operatively the patients will return for a follow up appointment along with their diary. If the patient does not have a follow-up appointment, the families may return the pain diary by email to the research coordinator or by mail with the given postage paid envelope. Demographic information such as age, race, gender, household income will be extracted from the diary and the electronic medical record. Information such as surgical technique, concurrent operations, post-operative pain prescription (types, weight based dosage, and total days prescribed) will be extracted from the electronic medical record and recorded as well. Outcomes measured will include pain scale rating and rates of complications between the two groups. We will also be investigating whether or not an opioid disposal pouch helps the process of disposing any leftover opioids from the trial. We will be providing all patients in the opioid arm an opioid disposal education document and randomizing half to receive the opioid disposal pouch.

Significance: If it can be demonstrated that non-opioid pain control after intracapsular adenotonsillectomy does not lead to increased pain or worse outcomes in certain pediatric age groups, a strong argument can be made for the cessation of opioid prescription for these ages following this technique. Given the widespread opioid epidemic, this would be a significant step in curbing the massive opioid problem, as well as reducing the adverse effects of opioid usage in pediatric populations.

ELIGIBILITY:
Inclusion Criteria:

• Patients age 3 - 17 undergoing adenotonsillectomy

Exclusion Criteria:

* Down syndrome
* History of coagulopathy
* Craniofacial abnormalities other than plagiocephaly or submucous cleft palate (SMCP)
* Caregivers who cannot speak, read, or write in English proficiently
* Patients who take opioids during the enrollment period
* Patients who take chronic opioids
* Pregnancy
* Allergy to or contraindication for taking any of the study medications
* Patients who have the inability to communicate
* Patients who have the inability to localize pain

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Chi, MD, Principal Investigator — Clinical Director, Division of Pediatric Otolaryngology, Children's Hospital of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Only co-investigators as listed under the University of Pittsburgh IRB (Institutional Review Board) protocol for this study will have access to all data and analysis. Data will be shared via UPMC-associated OneDrive and will only be shared between these investigators.

REFERENCES:
- [Background] Van Cleve WC, Grigg EB. Variability in opioid prescribing for children undergoing ambulatory surgery in the United States. J Clin Anesth. 2017 Sep;41:16-20. doi: 10.1016/j.jclinane.2017.05.014. Epub 2017 Jun 3. PMID 28802595
- [Background] Rudd RA, Seth P, David F, Scholl L. Increases in Drug and Opioid-Involved Overdose Deaths - United States, 2010-2015. MMWR Morb Mortal Wkly Rep. 2016 Dec 30;65(50-51):1445-1452. doi: 10.15585/mmwr.mm655051e1. PMID 28033313
- [Background] Schuchat A, Houry D, Guy GP Jr. New Data on Opioid Use and Prescribing in the United States. JAMA. 2017 Aug 1;318(5):425-426. doi: 10.1001/jama.2017.8913. No abstract available. PMID 28687823
- [Background] Feinberg AE, Chesney TR, Srikandarajah S, Acuna SA, McLeod RS; Best Practice in Surgery Group. Opioid Use After Discharge in Postoperative Patients: A Systematic Review. Ann Surg. 2018 Jun;267(6):1056-1062. doi: 10.1097/SLA.0000000000002591. PMID 29215370
- [Background] Monitto CL, Hsu A, Gao S, Vozzo PT, Park PS, Roter D, Yenokyan G, White ED, Kattail D, Edgeworth AE, Vasquenza KJ, Atwater SE, Shay JE, George JA, Vickers BA, Kost-Byerly S, Lee BH, Yaster M. Opioid Prescribing for the Treatment of Acute Pain in Children on Hospital Discharge. Anesth Analg. 2017 Dec;125(6):2113-2122. doi: 10.1213/ANE.0000000000002586. PMID 29189368
- [Background] Holte K, Kehlet H. Effect of postoperative epidural analgesia on surgical outcome. Minerva Anestesiol. 2002 Apr;68(4):157-61. PMID 12024074
- [Background] van Boekel RLM, Warle MC, Nielen RGC, Vissers KCP, van der Sande R, Bronkhorst EM, Lerou JGC, Steegers MAH. Relationship Between Postoperative Pain and Overall 30-Day Complications in a Broad Surgical Population: An Observational Study. Ann Surg. 2019 May;269(5):856-865. doi: 10.1097/SLA.0000000000002583. PMID 29135493
- [Background] Bean-Lijewski JD, Kruitbosch SH, Hutchinson L, Browne B. Post-tonsillectomy pain management in children: can we do better? Otolaryngol Head Neck Surg. 2007 Oct;137(4):545-51. doi: 10.1016/j.otohns.2007.06.731. PMID 17903568
- [Background] Luk LJ, Mosen D, MacArthur CJ, Grosz AH. Implementation of a Pediatric Posttonsillectomy Pain Protocol in a Large Group Practice. Otolaryngol Head Neck Surg. 2016 Apr;154(4):720-4. doi: 10.1177/0194599815627810. Epub 2016 Feb 16. PMID 26884362
- [Background] Kelly LE, Sommer DD, Ramakrishna J, Hoffbauer S, Arbab-Tafti S, Reid D, Maclean J, Koren G. Morphine or Ibuprofen for post-tonsillectomy analgesia: a randomized trial. Pediatrics. 2015 Feb;135(2):307-13. doi: 10.1542/peds.2014-1906. PMID 25624387

RESULTS

PARTICIPANT FLOW:
Groups:
- Opioid Pain Control: Patients in this group will be receiving triple therapy for pain control with oxycodone, acetaminophen, and ibuprofen. They will be asked to complete a pain diary which will be used to determine the level of pain control achieved with this regimen. A post-operative appointment between 4-8 weeks will be scheduled and the patient and caregiver will return the pain diary or by email/mail if no appointment was scheduled. The diary will be completed by post-operative day 14. Families will receive an opioid disposal education document.
Period: Overall Study
Arm/Group | Opioid Pain Control | Opioid Pain Control + Disposal Pouch | Non-opioid Pain Control
Started | 21 | 16 | 36
Completed | 13 | 8 | 24
Not Completed | 8 | 8 | 12
Not completed — Lost to Follow-up | 8 | 6 | 10
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Excludes patients withdrawn due to protocol violations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid Pain Control | Opioid Pain Control + Disposal Pouch | Non-opioid Pain Control | Total
Number analyzed (Participants) | 21 | 15 | 35 | 71
Age, Continuous [Median (Full Range); unit: years] | 4 [3 to 12] | 4 [3 to 8] | 4 [3 to 14] | 4 [3 to 14]
Age, Customized [Count of Participants; unit: Participants]
  3-7 years old | 18 | 13 | 31 | 62
  8-12 years old | 3 | 2 | 3 | 8
  13-17 years old | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14 | 28
  Male | 13 | 9 | 21 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 14 | 32 | 64
  Unknown or Not Reported | 3 | 1 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 3
  White | 19 | 14 | 30 | 63
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 21 | 15 | 35 | 71
BMI Centile [Median (Full Range); unit: percentile] | 72.31 [12.03 to 99.90] | 63.37 [6.67 to 94.28] | 72.50 [2.66 to 99.94] | 69.48 [2.66 to 99.94]

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Burden
Description: Average pain over 14 post-operative days before and after medications. This is quantified using the validated Wong-Baker FACES pain metric. The scale is from 0 to 10 with 10 being worse outcome. Patients receive a take-home pain diary and for 14 days report their maximum pain both before and after taking each pain medication. The mean of these pain ratings will be the primary outcome measure.
Time Frame: 14 days post-operatively
Population: Includes only patients who returned their pain diary (completed the study). Both those who did and did not receive the drug disposal bag are included in the opioid group, since this factor is not relevant to pain control. One patient in the opioid group reported no post-medication pain scores.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Number analyzed (Participants) | 21 | 24
score on a scale
  Before Medications | 3.2 [2.5 to 3.8] | 3.3 [2.6 to 4.1]
  After Medications: number analyzed (Participants) | 20 | 24
  After Medications | 1.1 [0.6 to 1.5] | 1.1 [0.6 to 1.5]
Statistical Analysis 1: Comparison: Opioid Pain Control vs Non-opioid Pain Control; Null hypothesis: No difference in average pain scores before medication between opioid and non-opioid groups; Test type: Superiority; p = 0.8, t-test, 2 sided
Statistical Analysis 2: Comparison: Opioid Pain Control vs Non-opioid Pain Control; Null hypothesis: No difference in average pain scores after medication between opioid and non-opioid groups; Test type: Superiority; p = 0.7, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: ED (Emergency Department) or Urgent Care Visits
Description: Number of emergency department or urgent care visits in 14 post-operative days - assessed via the electronic medical record and the take-home pain diary.
Time Frame: 14 days post-operatively
Population: Both those who did and did not receive the drug disposal bag are included in the opioid group, since this factor is not relevant to visiting the emergency room or urgent care. Excludes patients withdrawn due to protocol violations.
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Number analyzed (Participants) | 36 | 35
Participants
  0 ED or Urgent Care Visits | 36 | 33
  1 ED or Urgent Care Visit | 0 | 2
Statistical Analysis 1: Comparison: Opioid Pain Control vs Non-opioid Pain Control; Null hypothesis: There will be no difference in the proportion of patients visiting the emergency department or urgent care post-operatively between opioid and non-opioid groups; Test type: Superiority; p = 0.2, Fisher Exact

3. Other Pre Specified Outcome: Number of Readmissions
Description: Number of hospitalizations after discharge in 14 days - assessed using the electronic medical record and the take-home pain diary.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Frequency of Each Analgesic Used
Description: In the take-home pain diary, patients will place an 'x' on each time block every day that medication was given for each of the three medications. The frequencies will be summed for a total number and averaged within each group to determine the average number of times of each analgesic used.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Duration of Each Analgesic Used
Description: Using the results of the take-home pain diary, we will calculate the average number of days of use of each analgesic for each group. The last day after which there is no subsequent use of analgesic will define the end-point of the duration of use.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Pain Relief Satisfaction
Description: Score assigned by the patient at the end of 14 post-operative days in the take-home pain diary using a 5-point Likert scale of 0 (strongly disagree) to 4 (strongly agree). Patients will respond to the following statement "I am happy with the pain relief I received in the last 14 days" with responses ranging from strongly agree to strongly disagree. The responses will be assigned a numerical value and the average value for all subjects in the group will be reported as the overall pain relief satisfaction. Higher scores indicate a better outcome.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Post-operative Nursing Phone Calls
Description: Number of post-operative phone calls to nursing staff, obtained using the electronic medical record.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Night-time Awakenings
Description: Number of night-time awakenings reported in 14 days - assessed via the take-home pain diary.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Non-opioid Group Switching to Opioid Group
Description: Number of non-opioid group members switching to receiving opioid medication - assessed via the take-home pain diary.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Need for Follow-up Appointment
Description: Does the parent/guardian believe his/her child would require a follow-up appointment - assessed using the individual pain diary.
Time Frame: two months post-operatively
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Household Income
Description: Total household income ranges will be assessed in the take-home pain diary and reported.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Education Level
Description: Using the take-home pain diary, parents/guardians of the patients will identify the highest level of education achieved by anyone in the household.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Side Effects of Medications
Description: Number of any of the following side effects experienced: Nausea, vomiting, constipation, stomach ache, difficulty breathing. Assessed at follow-up and take-home pain diary.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Use of the Opioid Disposal Pouch
Description: Number of patients who reported that they used the opioid disposal pouch on the last page of the pain diary
Time Frame: Up until the return of the pain diary within 8 weeks of the surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5-9 weeks depending on the date of the follow-up appointment
Arm/Group | Opioid Pain Control | Opioid Pain Control + Disposal Pouch | Non-opioid Pain Control
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/16 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/16 | 1/36
Other Adverse Events (participants affected / at risk) | 3/21 | 1/16 | 2/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opioid Pain Control (N=21) | Opioid Pain Control + Disposal Pouch (N=16) | Non-opioid Pain Control (N=36)
Post-Tonsillectomy Hemorrhage Requiring Hospital Admission (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opioid Pain Control (N=21) | Opioid Pain Control + Disposal Pouch (N=16) | Non-opioid Pain Control (N=36)
Post-Tonsillectomy Hemorrhage Not Requiring Hospital Admission (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Decreased Oral Intake (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Emesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Eye/Cheek Edema (General disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to slow recruitment leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-16): https://cdn.clinicaltrials.gov/large-docs/61/NCT04791761/Prot_SAP_000.pdf